CLINICAL TRIAL: NCT07134829
Title: The Effects of Stroboscopic Visual Conditions on Gait and Lower Limb Muscle Activity in Individuals With Chronic Ankle Instability
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sahmyook University (Other)
Responsible Party: Principal Investigator, Suhyeon Jeong, Principal Investigator, MSc Candidate, Department of Physical Therapy, Sahmyook University, Sahmyook University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: SYU 2025-06-026-002
Record Dates: First submitted 2025-08-09; First posted 2025-08-21 (Actual); Last update posted 2025-08-21 (Actual); Status verified 2025-08

CONDITIONS: Chronic Ankle Instability
Keywords: Stroboscopic Glasses; Stroboscopic Vision; Gait Analysis; Surface Electromyography

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single Group - Chronic Ankle Instability (Experimental): All participants with chronic ankle instability will complete walking trials under three visual conditions: high-frequency stroboscopic glasses, low-frequency stroboscopic glasses, and no-glasses control. Each participant will perform three 5-meter walking trials per condition, with the order of conditions randomized.
  Interventions: Behavioral: Stroboscopic Visual Conditions

INTERVENTIONS:
Behavioral: Stroboscopic Visual Conditions — Participants will perform walking trials under three visual conditions: high-frequency stroboscopic glasses, low-frequency stroboscopic glasses, and no-glasses control. Each participant will complete three 5-meter walking trials per condition, with the order of conditions randomized. Gait parameters will be recorded using the GAITRite walkway system, and muscle activity will be measured using surface electromyography.

SUMMARY:
This interventional study will investigate the effects of stroboscopic visual conditions on gait patterns and lower limb muscle activation in adults with chronic ankle instability (CAI). CAI often results in impaired sensorimotor control, leading to altered gait strategies such as slower walking speed, shorter step length, and increased visual reliance. Stroboscopic glasses intermittently restrict visual input, potentially reducing visual dependence and enhancing proprioceptive feedback.

Participants will complete walking trials under three randomized visual conditions: high-frequency stroboscopic, low-frequency stroboscopic, and no-glasses control. Gait parameters will be measured using the GAITRite system, and surface electromyography (sEMG) will record activation of the tibialis anterior, peroneus longus, and gastrocnemius muscles. Findings may provide insight into sensorimotor adaptation mechanisms and inform rehabilitation strategies to improve functional stability in individuals with CAI.

DETAILED DESCRIPTION:
Chronic ankle instability (CAI) is a frequent outcome after ankle sprains, characterized by recurrent giving-way episodes, pain, and functional limitations. Approximately 40% of individuals with ankle sprains develop CAI, which is associated with deficits in proprioception, neuromuscular coordination, and postural stability. Increased visual reliance is a common compensatory strategy, but this can impair balance and gait when visual input is limited, raising the risk of re-injury.

Stroboscopic glasses alternate between transparent and opaque states, intermittently restricting visual information. This challenges the sensorimotor system, potentially reducing visual dependence and enhancing proprioceptive engagement. Prior research has shown benefits for static and dynamic balance, but little is known about effects on walking in CAI populations.

This randomized crossover study will assess the impact of high-frequency and low-frequency stroboscopic visual conditions compared with normal vision on gait and lower limb muscle activation in CAI. Adults aged 18-45 years with CAIT scores < 24 and a history of ankle instability within 6 months will be recruited. Exclusion criteria include recent lower limb surgery/fracture, systemic conditions affecting balance, or inability to follow instructions.

Participants will perform walking trials on a 5-meter GAITRite walkway under three randomized visual conditions:

1. High-frequency stroboscopic (rapid alternation)
2. Low-frequency stroboscopic (slower alternation)
3. No-glasses control (normal vision)

Gait parameters (step length, step time, gait velocity, swing/stance phases) will be measured, and sEMG (Noraxon) will assess activation of the tibialis anterior, peroneus longus, and gastrocnemius, normalized to MVIC. Subjective measures include CAIT, FAAM, IdFAI, and VAS pain scores.

It is hypothesized that stroboscopic conditions will produce measurable changes in gait and muscle activity compared with control, reflecting adaptive sensorimotor strategies that can inform rehabilitation programs to improve stability, mobility, and reduce re-injury risk.

ELIGIBILITY:
Inclusion Criteria:

* Individuals with a Cumberland Ankle Instability Tool (CAIT) score of less than 24
* Individuals diagnosed with ankle sprain or instability within the past 6 months

Exclusion Criteria:

* Individuals who have undergone lower limb surgery or experienced a fracture due to ankle trauma within the past 6 months
* Individuals with systemic diseases, such as cardiovascular disorders, that may affect balance
* Individuals who have difficulty understanding or following instructions during assessment or training

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 2025-08-31 (Estimated); Primary Completion 2025-09-28 (Estimated); Study Completion 2025-10-12 (Estimated)

PRIMARY OUTCOMES:
Change in Gait Velocity (cm/s) Under Different Stroboscopic Visual Conditions | Day 1 (single experimental session; immediately after each walking condition)
  Gait velocity will be measured using the GAITRite system under three visual conditions: high-frequency stroboscopic, low-frequency stroboscopic, and no stroboscopic. Each participant will perform three walking trials per condition over a 5-meter walkway. The average gait velocity (cm/s) will be calculated for each condition.

SECONDARY OUTCOMES:
Change in Step Length (cm) Under Different Stroboscopic Visual Conditions | Day 1 (single experimental session; immediately after each walking condition)
  Step length will be measured using the GAITRite system under three visual conditions. The average value (cm) will be calculated for each condition.
Change in Step Width (cm) Under Different Stroboscopic Visual Conditions | Day 1 (single experimental session; immediately after each walking condition)
  Step width will be measured using the GAITRite system under three visual conditions.
Change in Swing Phase (%) Under Different Stroboscopic Visual Conditions | Day 1 (single experimental session; immediately after each walking condition)
  Swing phase duration as a percentage of the gait cycle will be measured using the GAITRite system under three visual conditions.
Change in Single Limb Support (%) Under Different Stroboscopic Visual Conditions | Day 1 (single experimental session; immediately after each walking condition)
  Single limb support duration as a percentage of the gait cycle will be measured.
Change in Double Limb Support (%) Under Different Stroboscopic Visual Conditions | Day 1 (single experimental session; immediately after each walking condition)
  Double limb support duration as a percentage of the gait cycle will be measured.
Change in Tibialis Anterior Muscle Activation (%MVIC) Under Different Stroboscopic Visual Conditions | Day 1 (single experimental session; immediately after each walking condition)
  Surface electromyography (sEMG) will measure tibialis anterior muscle activation during walking. Data will be normalized to maximum voluntary isometric contraction (%MVIC).
Change in Peroneus Longus Muscle Activation (%MVIC) Under Different Stroboscopic Visual Conditions | Day 1 (single experimental session; immediately after each walking condition)
  sEMG will measure peroneus longus muscle activation during walking, normalized to %MVIC.
Change in Gastrocnemius Muscle Activation (%MVIC) Under Different Stroboscopic Visual Conditions | Day 1 (single experimental session; immediately after each walking condition)
  sEMG will measure gastrocnemius muscle activation during walking, normalized to %MVIC.
Correlation Between Foot and Ankle Ability Measure - ADL Subscale (FAAM-ADL) Score and Gait Velocity (cm/s) | Day 1 (questionnaire administered before walking tasks)
  Pearson's correlation will be computed between FAAM-ADL score (0-100; higher scores indicate better function) and gait velocity.
Correlation Between Foot and Ankle Ability Measure - Sports Subscale (FAAM-Sports) Score and Gait Velocity (cm/s) | Day 1 (questionnaire administered before walking tasks)
  Pearson's correlation will be computed between FAAM-Sports score (0-100; higher scores indicate better function) and gait velocity.
Correlation Between Identification of Functional Ankle Instability (IdFAI) Score and Gait Velocity (cm/s) | Day 1 (questionnaire administered before walking tasks)
  Pearson's correlation will be computed between IdFAI score (0-30; higher scores indicate greater instability) and gait velocity.
Correlation Between Visual Analogue Scale (VAS) Pain Score and Gait Velocity (cm/s) | Day 1 (questionnaire administered before walking tasks)
  Pearson's correlation will be computed between VAS pain score (0-10; higher scores indicate more severe pain) and gait velocity.

CONTACTS AND LOCATIONS:
Overall Officials: Seungwon Lee, PhD, Principal Investigator — Sahmyook University
Locations (1):
- Sahmyook University, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No